CLINICAL TRIAL: NCT01638000
Title: A Double-Blind, Randomized, Parallel Group, Multi-Centre Study to Evaluate the Efficacy and Safety of Mirabegron Compared to Solifenacin in Subjects With Overactive Bladder (OAB) Treated With Antimuscarinics and Dissatisfied Due to Lack of Efficacy
Brief Title: A Study to Evaluate the Efficacy and Safety of Mirabegron Compared to Solifenacin in Patients With Overactive Bladder Who Were Previously Treated With Another Medicine But Were Not Satisfied With That Treatment.
Acronym: BEYOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-EC-001; 2011-005713-37 (EudraCT Number)
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Urologic Diseases; Urinary Bladder, Overactive; Urinary Bladder Diseases
Keywords: Vesitrim; Frequency; Urgency; Urgency incontinence; Urinary incontinence; Overactive Bladder (OAB); Micturition; Mirabegron; YM178; Vesicare; Solifenacin
MeSH Terms: conditions — Urologic Diseases; Urinary Bladder, Overactive; Urinary Bladder Diseases; Urinary Incontinence | interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirabegron 50 mg (Experimental): Participants who received mirabegron 50 mg once daily for 12 weeks.
  Interventions: Drug: Mirabegron
- Solifenacin 5 mg (Active Comparator): Participants who received solifenacin 5 mg once daily for 12 weeks.
  Interventions: Drug: Solifenacin succinate

INTERVENTIONS:
Drug: Mirabegron — oral tablet
  Other Names: Betanis; YM178; Myrbetriq; Betmiga
  Arms: Mirabegron 50 mg
Drug: Solifenacin succinate — oral tablet
  Other Names: Vesicare; YM905; Vesikur; Vesitrim
  Arms: Solifenacin 5 mg

SUMMARY:
The purpose of the study was to assess the efficacy, safety and tolerability of mirabegron 50 mg versus (vs) solifenacin 5 mg in the treatment of patients with OAB who were dissatisfied with their treatment due to lack of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to complete the micturition diary and questionnaires correctly
* Subject has symptoms of OAB (urinary frequency and urgency with or without urgency incontinence) for at least 3 months
* Subject is currently or has previously received at least one antimuscarinic agent intended to treat their OAB. The last antimuscarinic must have been taken for at least 4 weeks and taken within 6 months prior to the Screening Visit

Exclusion Criteria:

* Female subject is breastfeeding, pregnant, intends to become pregnant during the study, or of childbearing potential is sexually active and not practicing a highly reliable method of birth control
* Subject has neurogenic bladder
* Subject has significant stress incontinence or mixed stress/urgency incontinence where stress is the predominant factor as determined by the investigator (for female subjects confirmed by a cough provocation test)
* Subject has an indwelling catheter or practices intermittent self-catheterization
* Subject has diabetic neuropathy
* Subject has evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs
* Subject has uncontrolled narrow angle glaucoma, urinary or gastric retention, severe ulcerative colitis, toxic megacolon, myasthenia gravis or any other medical condition which makes the use of anticholinergics contraindicated
* The subject is currently receiving or has a history of treatment with intravesical botulinum toxin (cosmetic use is acceptable) or resiniferatoxin within 9 months prior to screening
* Subject receives non-drug treatment including electro-stimulation therapy (with the exception of a bladder training program or pelvic floor exercises which started more than 30 days prior to screening)
* Subject has moderate to severe hepatic impairment
* Subject has severe renal impairment or end stage renal disease
* Subject has severe uncontrolled hypertension
* Subject has a clinically significant abnormal electrocardiogram (ECG) or has a known history of QT prolongation or currently taking medication known to prolong the QT interval
* Subject has a known or suspected hypersensitivity to solifenacin, mirabegron or any of the inactive ingredients
* Subject has a concurrent malignancy or history of cancer (except noninvasive skin cancer) within the last 5 years prior to screening
* Subject has been treated with an experimental device within 30 days or received an experimental agent within the longer of 30 days or five half-lives
* Subject is using prohibited medications which cannot be stopped safely at the Screening Visit. Subject is excluded if using restricted medications not meeting protocol-specified criteria
* Subject's last antimuscarinic treatment was solifenacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1887 (Actual)
Dates: Start 2012-06-12 (Actual); Primary Completion 2013-04-24 (Actual); Study Completion 2013-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe Ltd.
Locations (217):
- Armenia (5):
  - Site: 37406, Yerevan
  - Site: 37404, Yerevan
  - Site: 37403, Yerevan
  - Site: 37401, Yerevan
  - Site: 37402, Yerevan
- Austria (8):
  - Site: 43006, Baden
  - Site: 43014, Graz
  - Site: 43015, Innsbruck
  - Site: 43013, Linz
  - Site: 43005, Oberwart
  - Site: 43011, Vienna
  - Site: 43002, Vienna
  - Site: 43003, Wels
- Belarus (3):
  - Site: 37502, Minsk
  - Site: 37501, Minsk
  - Site: 37504, Vitebsk
- Belgium (6):
  - Site: 32006, Brussels
  - Site: 32008, Deurne
  - Site: 32001, Edegem
  - Site: 32004, Ghent
  - Site: 32007, Leuven
  - Site: 32005, Liège
- Bulgaria (7):
  - Site: 35902, Burgas
  - Site: 35909, Haskovo
  - Site: 35901, Lovech
  - Site: 35905, Plovdiv
  - Site: 35906, Sofia
  - Site: 35908, Sofia
  - Site: 35903, Sofia
- Canada (10):
  - Site: 10010, Abbotsford
  - Site: 10011, Barrie
  - Site: 10001, Bathurst
  - Site: 10003, Brampton
  - Site: 10005, Brantford
  - Site: 10007, Kingston
  - Site: 10002, Montreal
  - Site: 10009, Sherbrooke
  - Site: 10004, Toronto
  - Site: 10008, Victoria
- Czechia (8):
  - Site: 42004, Bohumín
  - Site: 42003, Brno
  - Site: 42001, Hradec Králové
  - Site: 42002, Jihlava
  - Site: 42006, Plzen-Lochotin
  - Site: 42005, Prague
  - Site: 42008, Prague
  - Site: 42007, Prague
- Denmark (5):
  - Site: 45002, Aalborg
  - Site: 45001, Aarhus N
  - Site: 45005, Frederiksbjerg
  - Site: 45004, Hvidovre
  - Site: 45003, Odense C
- Finland (3):
  - Site: 35802, Jyväskylä
  - Site: 35801, Oulu
  - Site: 35804, Tampere
- France (13):
  - Site: 33010, Angers
  - Site: 33007, Colmar
  - Site: 33011, Dijon
  - Site: 33002, Marseille
  - Site: 33006, Marseille
  - Site: 33013, Nîmes
  - Site: 33004, Orléans
  - Site: 33001, Paris
  - Site: 33005, Paris
  - Site: 33003, Rouen
  - Site: 33014, Suresnes
  - Site: 33017, Tours
  - Site: 33015, Valence
- Georgia (3):
  - Site: 99501, Tbilisi
  - Site: 99502, Tbilisi
  - Site: 99503, Tbilisi
- Germany (2):
  - Site: 49006, Bad Ems
  - Site: 49009, Halle
- Greece (9):
  - Site: 30005, Alexandroupoli
  - Site: 30009, Athens
  - Site: 30007, Athens
  - Site: 30001, Athens
  - Site: 30006, Heraklion
  - Site: 30008, Larissa
  - Site: 30004, Pátrai
  - Site: 30010, Thessaloniki
  - Site: 30002, Thessaloniki
- Hungary (6):
  - Site: 36003, Budapest
  - Site: 36004, Budapest
  - Site: 36005, Csongrád
  - Site: 36006, Nyíregyháza
  - Site: 36001, Salgótarján
  - Site: 36002, Szekszárd
- Ireland (6):
  - Site: 35304, Cork
  - Site: 35302, Dublin
  - Site: 35306, Dublin
  - Site: 35301, Dublin
  - Site: 35303, Tralee
  - Site: 35305, Waterford
- Italy (8):
  - Site: 39001, Avellino
  - Site: 39005, Catanzaro
  - Site: 39003, Cinisello Balsamo
  - Site: 39002, Florence
  - Site: 39008, Milan
  - Site: 39010, Pavia
  - Site: 39006, Perugia
  - Site: 39007, Treviglio
- Kazakhstan (4):
  - Site: 77705, Almaty
  - Site: 77706, Almaty
  - Site: 77703, Astana
  - Site: 77702, Astana
- Latvia (3):
  - Site: 37103, Liepāja
  - Site: 37102, Riga
  - Site: 37101, Riga
- Lebanon (2):
  - Site: 96102, Byblos
  - Site: 96103, El Achrafiyé
- Lithuania (2):
  - Site: 37001, Kaunas
  - Site: 37003, Vilnius
- Netherlands (7):
  - Site: 31010, Amsterdam
  - Site: 31005, Eindhoven
  - Site: 31004, Enschede
  - Site: 31007, Nijmegen
  - Site: 31001, Tilburg
  - Site: 31008, Utrecht
  - Site: 31006, Zwolle
- Norway (3):
  - Site: 47002, Hamar
  - Site: 47005, Trondheim
  - Site: 47001, Tønsberg
- Poland (6):
  - Site: 48007, Kolbuszowa Dolna
  - Site: 48006, Krakow
  - Site: 48001, Lublin
  - Site: 48004, Piaseczno
  - Site: 48003, Warsaw
  - Site: 48005, Wroclaw
- Portugal (5):
  - Site: 35105, Lisbon
  - Site: 35104, Lisbon
  - Site: 35102, Matosinhos Municipality
  - Site: 35103, Porto
  - Site: 35101, Setúbal
- Russia (13):
  - Site: 70007, Moscow
  - Site: 70001, Moscow
  - Site: 70008, Moscow
  - Site: 70005, Moscow
  - Site: 70006, Moscow
  - Site: 70011, Moscow
  - Site: 70002, Moscow
  - Site: 70003, Moscow
  - Site: 70013, Saint Petersburg
  - Site: 70012, Saint Petersburg
  - Site: 70004, Saint Petersburg
  - Site: 70010, Saint Petersburg
  - Site: 70009, Saint Petersburg
- Slovakia (6):
  - Site: 42104, Galanta
  - Site: 42106, Martin
  - Site: 42103, Piešťany
  - Site: 42101, Poprad
  - Site: 42105, Trenčín
  - Site: 42102, Žilina
- Slovenia (5):
  - Site: 38603, Ljubljana
  - Site: 38604, Ljubljana
  - Site: 38601, Maribor
  - Site: 38602, Maribor
  - Site: 38606, Novo Mesto
- Spain (11):
  - Site: 34001, Barcelona
  - Site: 34002, Barcelona
  - Site: 34009, Bilbao
  - Site: 34010, Donostia / San Sebastian
  - Site: 34004, Madrid
  - Site: 34005, Madrid
  - Site: 34003, Madrid
  - Site: 34011, Mendaro
  - Site: 34013, Murcia
  - Site: 34014, Seville
  - Site: 34012, Valencia
- Sweden (7):
  - Site: 46007, Gothenburg
  - Site: 46004, Halmstad
  - Site: 46005, Karlshamn
  - Site: 46003, Norrtälje
  - Site: 46002, Stockholm
  - Site: 46001, Stockholm
  - Site: 46006, Uppsala
- Switzerland (2):
  - Site: 41001, Frauenfeld
  - Site: 41003, Zurich
- Turkey (Türkiye) (9):
  - Site: 90005, Ankara
  - Site: 90003, Ankara
  - Site: 90011, Denizli
  - Site: 90007, Diyarbakır
  - Site: 90004, Istanbul
  - Site: 90001, Izmir
  - Site: 90008, Izmir
  - Site: 90009, Manisa
  - Site: 90010, Sivas
- Ukraine (5):
  - Site: 38007, Chernivtsi
  - Site: 38004, Dnipro
  - Site: 38001, Kharkiv
  - Site: 38002, Kiev
  - Site: 38003, Lviv
- United Kingdom (25):
  - Site: 44027, Aberdeen
  - Site: 44029, Birmingham
  - Site: 44025, Cambridge
  - Site: 44030, Chichester
  - Site: 44028, Croydon
  - Site: 44003, Devon
  - Site: 44001, Edgbaston
  - Site: 44011, Glasgow
  - Site: 44023, Harrow
  - Site: 44006, Kent
  - Site: 44012, Leeds
  - Site: 44019, Leicester
  - Site: 44008, Liverpool
  - Site: 44010, London
  - Site: 44017, London
  - Site: 44013, Newcastle upon Tyne
  - Site: 44022, Northwood
  - Site: 44021, Nottingham
  - Site: 44009, Plymouth
  - Site: 44007, Reading
  - Site: 44005, Sheffield
  - Site: 44020, Southampton
  - Site: 44026, Taunton
  - Site: 44024, West Yorkshire
  - Site: 44002, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=27

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited for this study were men and women with overactive bladder (OAB) who had received 1 or more antimuscarinics in the past and who were dissatisfied with their last antimuscarinic treatment due to lack of efficacy (provided that their previous antimuscarinic was not solifenacin).
Pre-assignment Details: Participants entered a 2-week, single-blind, placebo run-in period and completed a daily diary (including 3 consecutive days prior to the randomization visit for micturition and incontinence). After this, participants' eligibility criteria were re-confirmed and they were then randomized into the double-blind treatment period of the study.
Period: Overall Study
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Started | 943 | 944
Received at Least 1 Double-Blind Dose | 936 | 934
Completed | 883 | 873
Not Completed | 60 | 71
Not completed — Randomized but Never Received Drug | 7 | 10
Not completed — Adverse Event | 14 | 16
Not completed — Lack of Efficacy | 5 | 6
Not completed — Protocol Violation | 11 | 13
Not completed — Withdrawal by Subject | 21 | 24
Not completed — Miscellaneous | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) - consisted of all randomized patients who received ≥ 1 dose of double-blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg | Total
Number analyzed (Participants) | 936 | 934 | 1870
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (14.25) | 57.4 (13.60) | 57.0 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 712 | 709 | 1421
  Male | 224 | 225 | 449
Mean Micturitions / 24 hours [Mean (Standard Deviation); unit: micturitions] — SAF population. The number of participants are 933 and 932. A micturition is any voluntary urination (excluding incontinence only episodes). The mean number of micturitions per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
  micturitions | 11.6 (3.25) | 11.4 (2.89) | 11.5 (3.08)
Mean Incontinence Episodes / 24 hours [Mean (Standard Deviation); unit: incontinence episodes] — SAF population with baseline value > 0. The number of participants are 410 and 424. An incontinence episode is any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
  incontinence episodes | 2.1 (2.30) | 2.1 (2.05) | 2.1 (2.17)
Mean Urgency Incontinence Episodes / 24 hours [Mean (Standard Deviation); unit: urgency incontinence episodes] — SAF population with baseline value > 0. The number of participants are 401 and 413. An urgency incontinence episode is any involuntary leakage of urine accompanied by or immediately proceeded by urgency. The mean number of urgency incontinence episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
  urgency incontinence episodes | 1.9 (1.99) | 2.0 (1.94) | 2.0 (1.96)
Mean Urgency Episodes (grade 3 or 4) / 24 hours [Mean (Standard Deviation); unit: urgency episodes] — SAF population with baseline value > 0. The number of participants are 931 and 931. An urgency episode is a sudden compelling desire to pass urine immediately followed by an incontinent event or the patient having to rush to the toilet and make it in time; severity recorded as 3 (severe urgency) or 4 (urgency incontinence) on the Patient Perception of the Intensity of Urgency Scale (PPIUS) validated scale. The mean number of urgency episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
  urgency episodes | 7.7 (4.75) | 7.8 (4.46) | 7.8 (4.61)
Mean Level of Urgency [Mean (Standard Deviation); unit: units on a scale] — SAF population. The number of participants are 933 and 932. Urgency level was rated by the participant during the 3-day micturition diary period using the PPIUS 5-point categorical scale: 0. No urgency; 1. Mild urgency; 2. Moderate urgency; 3. Severe urgency; 4. Urgency incontinence.
  units on a scale | 2.6 (0.49) | 2.6 (0.49) | 2.6 (0.49)
Mean Nocturia Episodes / 24 hours [Mean (Standard Deviation); unit: nocturia episodes] — SAF population with baseline value > 0. The number of participants are 890 and 895. A nocturia episode is defined as waking at night ≥ 1 times to void (i.e., any voiding associated with sleep disturbance between the time the patient goes to bed with the intention to sleep until the time the patient gets up in the morning with the intention to stay awake). The mean number of nocturia episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
  nocturia episodes | 2.3 (1.41) | 2.3 (1.42) | 2.3 (1.41)
Mean Number of Pads Used / 24 hours [Mean (Standard Deviation); unit: pads] — SAF population with baseline value > 0. The number of participants are 585 and 580. The mean number of pads per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
  pads | 3.1 (3.43) | 3.3 (3.70) | 3.2 (3.57)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Final Visit in the Mean Number of Micturitions Per 24 Hours
Description: A micturition is any voluntary urination (excluding incontinence only episodes). The mean number of micturitions per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
Time Frame: Baseline and final visit (up to Week 12)
Population: Per Protocol Set (PPS) - all randomized participants who took ≥1 dose of double-blind study drug and who recorded ≥1 micturition in the baseline diary and ≥1 micturition in a post-baseline diary who had completed the study with no major protocol violations which could impact the primary endpoint. Last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 865 | 853
micturitions | -2.95 (0.087) | -3.13 (0.088)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; The non-inferiority of mirabegron vs. solifencacin on the change from baseline to final visit in the mean number of micturitions per 24 hours; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the lower limit of the 95% CI for difference of adjusted change from baseline between solifenacin 5 mg and mirabegron 50 mg was > -0.20. Differences of adjusted means were calculated by subtracting the adjusted mean of mirabegron 50 mg from the adjusted mean of solifenacin 5 mg. Overall power calculation was 80% for a 1-sided test and significance level of 0.025; p = 0.15, ANCOVA — If p<0.05, this indicated superiority in favor of the treatment group with the largest improvement at specified visit; Treatment group, gender, age group (<65, ≥65), number of prior antimuscarinics (1, ≥2), geographic region as fixed factors and baseline as a covariate; least squares mean difference = -0.18, 95% CI 2-sided [-0.42 to 0.06], Standard Error of Mean 0.124

2. Secondary Outcome: Percentage of Participants Reporting at Least One Treatment-emergent Adverse Event of Dry Mouth, Constipation or Blurred Vision During Double-blind Treatment Period
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE; defined as any untoward medical occurrence in a patient administered a study drug) that started or worsened in the period from the first double-blind medication intake until 30 days after the last double-blind medication intake. The following TEAEs were selected for inclusion in the analysis: Dry mouth (aptyalism, dry mouth, dry throat), constipation (constipation), blurred vision (vision blurred, myopia, refraction disorder, accommodation disorder).
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 16 weeks)
Population: SAF population
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 936 | 934
percentage of participants
  Overall | 5 | 7.4
  Dry mouth | 3.1 | 5.8
  Dry throat | 0.1 | 0.1
  Blurred vision | 0.6 | 0.4
  Constipation | 2.2 | 2.5
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Difference vs Mirabegron. Differences of the percentages were calculated by subtracting the percentage of mirabegron 50 mg group from the percentage of solifenacin 5 mg group; Test type: Superiority or Other; p = 0.030, Regression, Logistic — If P <0.05, this indicates superiority in favor of the treatment group with the smallest percentage of participants with at least 1 TEAE of dry mouth, constipation or blurred vision during the double-blind period at the final visit; Included treatment group, sex, age group (< 65, ≥ 65), number of prior antimuscarinics (1, ≥ 2) and geographic region as factors; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.04 to 2.25]

3. Secondary Outcome: Change From Baseline to 4, 8 and 12 Weeks of Treatment in Mean Number of Micturitions Per 24 Hours
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: Full Analysis Set (FAS) - consisted of all randomized participants who took ≥ 1 dose of double-blind study drug and who recorded ≥1 micturition measurement in the baseline diary and ≥1 micturition measurement in a post-baseline diary. N is the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
micturitions
  Week 4 [N=916,906] | -2.37 (0.083) | -2.33 (0.083)
  Week 8 [N=888,876] | -2.77 (0.084) | -3.00 (0.085)
  Week 12 [N=870,856] | -3.02 (0.088) | -3.21 (0.089)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Difference vs. Mirabegron. Differences of adjusted means were calculated by subtracting the adjusted mean of mirabegron 50 mg from the adjusted mean of solifenacin 5 mg; Test type: Superiority or Other; p = 0.71, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; least squares mean difference = 0.04, 95% CI 2-sided [-0.19 to 0.27], Standard Error of Mean 0.117
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Difference vs. Mirabegron. Differences of adjusted means were calculated by subtracting the adjusted mean of mirabegron 50 mg from the adjusted mean of solifenacin 5 mg; Test type: Superiority or Other; p = 0.053, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; least squares mean difference = -0.23, 95% CI 2-sided [-0.47 to 0.00], Standard Error of Mean 0.119
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Difference vs. Mirabegron. Differences of adjusted means were calculated by subtracting the adjusted mean of mirabegron 50 mg from the adjusted mean of solifenacin 5 mg; Test type: Superiority or Other; p = 0.12, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; least squares mean difference = -0.20, 95% CI 2-sided [-0.44 to 0.05], Standard Error of Mean 0.125

4. Secondary Outcome: Number of Incontinence Episodes at 4, 8 and 12 Weeks of Treatment and at the Final Visit
Description: An incontinence episode is any involuntary leakage of urine. The total number of incontinence episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period prior to each visit.
Time Frame: Week 4, Week 8, Week 12
Population: FAS-Incontinence (FAS-I) - consisted of all FAS participants with ≥1 incontinence episode at baseline. LOCF was used for final visit only. N is the number of participants with available data at each time point.
Measure: Mean (Standard Error); unit: incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 405 | 413
incontinence episodes
  Week 4 [N=404,410] | 2.64 (0.280) | 2.25 (0.217)
  Week 8 [N=387,397] | 2.19 (0.457) | 1.28 (0.135)
  Week 12 [N=381,387] | 2.07 (0.562) | 1.08 (0.124)
  Final visit [N=404,413] | 2.13 (0.533) | 1.29 (0.157)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.33, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; Treatment group, gender, age group (<65, ≥65), number of prior antimuscarinics (1, ≥2), geographic region and baseline as covariates; Rate ratio = 0.90, 95% CI 2-sided [0.73 to 1.11]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.21, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 0.84, 95% CI 2-sided [0.64 to 1.10]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.83, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 0.97, 95% CI 2-sided [0.71 to 1.32]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final Visit Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.57, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; Treatment group, gender, age group (<65,≥ 65), number of prior antimuscarinics (1, ≥2), geographic region and baseline as covariates; Rate ratio = 0.92, 95% CI 2-sided [0.68 to 1.24]

5. Secondary Outcome: Change From Baseline to 4, 8 and 12 Weeks of Treatment in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode is any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: FAS-I population. N is the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 405 | 413
incontinence episodes
  Week 4 [N=404,410] | -1.22 (0.063) | -1.30 (0.063)
  Week 8 [N=387,397] | -1.37 (0.093) | -1.59 (0.092)
  Week 12 [N=381,387] | -1.41 (0.115) | -1.66 (0.114)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.36, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; From stratified rank ANCOVA analysis; Least squares mean difference = -0.08, 95% CI 2-sided [-0.25 to 0.10], Standard Error of Mean 0.089
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.12, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; From the stratified rank ANCOVA analysis; Least squares mean difference = -0.22, 95% CI 2-sided [-0.48 to 0.03], Standard Error of Mean 0.130
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Difference vs. Mirabegron. Difference of the adjusted mean is calculated by subtracting the adjusted mean of mirabegron from the adjusted mean of solifenacin; Test type: Superiority or Other; p = 0.47, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; From the stratified rank ANCOVA analysis; Least squares mean difference = -0.25, 95% CI 2-sided [-0.57 to 0.07], Standard Error of Mean 0.163

6. Secondary Outcome: Number of Urgency Incontinence Episodes at 4, 8 and 12 Weeks of Treatment and at the Final Visit
Description: An urgency incontinence episode is any involuntary leakage of urine accompanied by or immediately proceeded by urgency. The total number of urgency incontinence episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period prior to each visit.
Time Frame: Week 4, Week 8, Week 12
Population: FAS-I population. LOCF was used for final visit only. Only participants with at least one urgency incontinence episode at baseline were included in the analysis. N is the number of participants with available data at each time point.
Measure: Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 405 | 413
urgency incontinence episodes
  Week 4 [N=395,399] | 2.27 (0.230) | 2.16 (0.213)
  Week 8 [N=379,386] | 1.74 (0.227) | 1.13 (0.125)
  Week 12 [N=373,377] | 1.44 (0.217) | 1.03 (0.120)
  Final visit [N=395,402] | 1.51 (0.211) | 1.23 (0.150)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.44, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 0.92, 95% CI 2-sided [0.74 to 1.14]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.11, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 0.79, 95% CI 2-sided [0.60 to 1.06]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.78, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.05, 95% CI 2-sided [0.76 to 1.45]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final Visit Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.85, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 0.97, 95% CI 2-sided [0.71 to 1.33]

7. Secondary Outcome: Change From Baseline to 4, 8 and 12 Weeks of Treatment in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: An urgency incontinence episode is any involuntary leakage of urine accompanied by or immediately proceeded by urgency. The mean number of urgency incontinence episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: FAS-I population. Only participants with at least one urgency incontinence episode at baseline were included in the analysis. N is the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 405 | 413
urgency incontinence episodes
  Week 4 [N=395,399] | -1.22 (0.057) | -1.24 (0.057)
  Week 8 [N=379,386] | -1.39 (0.050) | -1.56 (0.050)
  Week 12 [N=373,377] | -1.49 (0.047) | -1.59 (0.047)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.66, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; From stratified rank ANCOVA analysis; Least squares mean difference = -0.02, 95% CI 2-sided [-0.18 to 0.14], Standard Error of Mean 0.081
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.17, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; From the stratified rank ANCOVA analysis; Least squares mean difference = -0.17, 95% CI 2-sided [-0.31 to -0.03], Standard Error of Mean 0.070
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.66, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; From the stratified rank ANCOVA analysis; Least squares mean difference = -0.11, 95% CI 2-sided [-0.24 to 0.02], Standard Error of Mean 0.066

8. Secondary Outcome: Change From Baseline to 4, 8 and 12 Weeks of Treatment and at the Final Visit in Mean Number of Urgency Episodes (Grade 3 or 4) Per 24 Hours
Description: An urgency episode is a sudden compelling desire to pass urine immediately followed by an incontinent event or the patient having to rush to the toilet and make it in time; severity recorded as 3 (severe urgency) or 4 (urgency incontinence) on the Patient Perception of the Intensity of Urgency Scale (PPIUS) validated scale. The mean number of urgency episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: FAS population. LOCF was used for final visit only. Only participants with at least one urgency episode (grade 3 or 4) at baseline were included in this analysis. N is the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
urgency episodes
  Week 4 [N=915,905] | -3.75 (0.113) | -3.88 (0.114)
  Week 8 [N=887,875] | -4.44 (0.111) | -4.79 (0.112)
  Week 12 [N=869,855] | -4.67 (0.116) | -4.99 (0.117)
  Final Visit [N=919,909] | -4.61 (0.115) | -4.84 (0.115)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.43, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.13, 95% CI 2-sided [-0.44 to 0.19], Standard Error of Mean 0.160
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.027, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.35, 95% CI 2-sided [-0.66 to -0.04], Standard Error of Mean 0.157
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.053, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.32, 95% CI 2-sided [-0.64 to 0.00], Standard Error of Mean 0.164
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final Visit Difference vs. Mirabegron. Differences of adjusted means were calculated by subtracting the adjusted mean of mirabegron 50 mg from the adjusted mean of solifenacin 5 mg; Test type: Superiority or Other; p = 0.16, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.23, 95% CI 2-sided [-0.55 to 0.09], Standard Error of Mean 0.163

9. Secondary Outcome: Change From Baseline to 4, 8 and 12 Weeks of Treatment and at the Final Visit in Mean Level of Urgency
Description: Urgency level was rated by the participant during the 3-day micturition diary period using the PPIUS 5-point categorical scale: 0. No urgency; 1. Mild urgency; 2. Moderate urgency; 3. Severe urgency; 4. Urgency incontinence.
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: FAS population. LOCF was used in final visit only. N is the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
units on a scale
  Week 4 [N=916,906] | -0.36 (0.016) | -0.36 (0.017)
  Week 8 [N=888,876] | -0.50 (0.019) | -0.52 (0.019)
  Week 12 [N=870,856] | -0.60 (0.023) | -0.60 (0.023)
  Final visit [N=920,910] | -0.58 (0.022) | -0.57 (0.022)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.99, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.023
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.47, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.02, 95% CI 2-sided [-0.07 to 0.03], Standard Error of Mean 0.027
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.99, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.00, 95% CI 2-sided [-0.06 to 0.06], Standard Error of Mean 0.032
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.74, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.01, 95% CI 2-sided [-0.05 to 0.07], Standard Error of Mean 0.031

10. Secondary Outcome: Number of Pads Used at 4, 8 and 12 Weeks of Treatment and at the Final Visit
Description: The total number of pads per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period prior to each visit.
Time Frame: Week 4, Week 8, Week 12
Population: FAS population. LOCF was used in final visit only. Only participants with at least one pad used at baseline were included in this analysis. N is the number of participants with available data at each time point.
Measure: Mean (Standard Error); unit: pads
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
pads
  Week 4 [N=574,563] | 4.25 (0.324) | 4.26 (0.297)
  Week 8 [N=551,543] | 3.33 (0.284) | 3.27 (0.236)
  Week 12 [N=543,532] | 3.19 (0.304) | 3.04 (0.244)
  Final visit [N=576,565] | 3.32 (0.300) | 3.19 (0.248)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.67, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.03, 95% CI 2-sided [0.89 to 1.20]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.073, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.17, 95% CI 2-sided [0.99 to 1.39]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.25, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.12, 95% CI 2-sided [0.92 to 1.37]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final Visit Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.40, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.08, 95% CI 2-sided [0.90 to 1.31]

11. Secondary Outcome: Change From Baseline in Mean Number of Pads Used Per 24 Hours After 4, 8 and 12 Weeks of Treatment
Description: The mean number of pads per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
Time Frame: Baseline and Week 4, Week 8 , Week 12
Population: FAS population. Only participants with at least one pad used at baseline were included in this analysis. N is the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
pads
  Week 4 [M=574,563] | -1.80 (0.081) | -1.82 (0.081)
  Week 8 [N=551,543] | -2.10 (0.070) | -2.14 (0.070)
  Week 12 [N=543,532] | -2.14 (0.078) | -2.20 (0.079)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.84, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.02, 95% CI 2-sided [-0.25 to 0.20], Standard Error of Mean 0.115
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.63, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.05, 95% CI 2-sided [-0.24 to 0.15], Standard Error of Mean 0.099
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.59, ANCOVA — if p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.06, 95% CI 2-sided [-0.28 to 0.16], Standard Error of Mean 0.111

12. Secondary Outcome: Number of Nocturia Episodes at 4, 8 and 12 Weeks of Treatment and at the Final Visit
Description: A nocturia episode is defined as waking at night ≥1 times to void (i.e., any voiding associated with sleep disturbance between the time the patient goes to bed with the intention to sleep until the time the patient gets up in the morning with the intention to stay awake). The total number of nocturia episodes were calculated from the data recorded by the participant during the 3-day micturition diary period prior to each visit.
Time Frame: Week 4, Week 8, Week 12
Population: FAS population. LOCF was used for final visit only. Only participants with at least one nocturia episode at baseline were included in the analysis. N is the number of participants with available data at each time point.
Measure: Mean (Standard Error); unit: nocturia episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
nocturia episodes
  Week 4 [N=877,871] | 4.78 (0.120) | 5.12 (0.139)
  Week 8 [N=850, 844] | 4.26 (0.118) | 4.41 (0.117)
  Week 12 [N=831,828] | 3.94 (0.115) | 4.06 (0.116)
  Final Visit [N=879,875] | 4.05 (0.120) | 4.13 (0.114)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.068, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.05, 95% CI 2-sided [1.00 to 1.11]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.21, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.04, 95% CI 2-sided [0.98 to 1.11]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.52, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.02, 95% CI 2-sided [0.95 to 1.10]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final Visit Rate Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.44, Poisson regression — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 4, analysis 1]; Rate ratio = 1.03, 95% CI 2-sided [0.96 to 1.10]

13. Secondary Outcome: Change From Baseline in Mean Number of Nocturia Episodes Per 24 Hours After 4, 8 and 12 Weeks of Treatment
Description: A nocturia episode is defined as waking at night ≥1 times to void (i.e., any voiding associated with sleep disturbance between the time the patient goes to bed with the intention to sleep until the time the patient gets up in the morning with the intention to stay awake). The mean number of nocturia episodes per 24 hours were calculated from the data recorded by the participant during the 3-day micturition diary period.
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: FAS population. Only participants with at least one nocturia episode at baseline were included in the analysis. N is the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
nocturia episodes
  Week 4 [N=877,871] | -0.72 (0.033) | -0.63 (0.034)
  Week 8 [N=850,844] | -0.90 (0.031) | -0.87 (0.031)
  Week 12 [N=831,828] | -0.98 (0.032) | -0.97 (0.033)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.058, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.09, 95% CI 2-sided [-0.00 to 0.18], Standard Error of Mean 0.047
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.50, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.03, 95% CI 2-sided [-0.06 to 0.12], Standard Error of Mean 0.044
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.81, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.01, 95% CI 2-sided [-0.08 to 0.10], Standard Error of Mean 0.046

14. Secondary Outcome: Percentage of Participants With Normalization of Micturitions at Weeks 4, 8, 12 and Final Visit
Description: A responder is defined as a participant who has ≥8 micturitions at baseline and has <8 micturitions per 24 hours during the treatment period at each specified visit, where change from baseline is <0.
Time Frame: Week 4, Week 8, Week 12
Population: FAS population. LOCF was used for final visit only. N is the number of participants with available data at each timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
percentage of participants
  Week 4 [N=916,906] | 32.3 | 33.9
  Week 8 [N=888,876] | 41.2 | 46.9
  Week 12 [N=870,856] | 44.8 | 49.3
  Final visit [N=920,910] | 44.2 | 48.8
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Odds ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.67, Regression, Logistic — If p<0.05, this indicates superiority in favor of the treatment group with the largest percentage of responders at specified visit; Treatment group, gender, age group (<65,≥ 65), number of prior antimuscarinics (1, ≥2), geographic region and baseline value as factors; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.85 to 1.28]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Odds ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.026, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.03 to 1.53]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Odds ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.11, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.97 to 1.44]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final Visit Odds ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.093, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.97 to 1.43]

15. Secondary Outcome: Percentage of Participants With 50% Reduction in Incontinence Episodes at Weeks 4, 8, 12 and Final Visit
Description: A responder is defined as a participant with at least 50% decrease from baseline in mean number of incontinence episodes per 24 hours during the treatment period at specified visit.
Time Frame: Week 4, Week 8, Week 12
Population: FAS-I population. LOCF was used for final visit only. N is the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 405 | 413
percentage of participants
  Week 4 [N=404,410] | 75.5 | 77.3
  Week 8 [N=387,397] | 85.5 | 86.9
  Week 12 [N=381,387] | 86.1 | 89.1
  Final visit [N=404,413] | 85.1 | 88.1
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.74, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.76 to 1.48]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.74, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.71 to 1.63]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.29, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.81 to 2.00]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.29, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.82 to 1.90]

16. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes at Weeks 4, 8, 12 and Final Visit
Description: A responder is defined as a participant who reported incontinence episodes at baseline and reported no incontinence episodes during the treatment period at specified visit.
Time Frame: Week 4, Week 8, Week 12
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 405 | 413
percentage of participants
  Week 4 [N=404,410] | 47.3 | 52.0
  Week 8 [N=387,397] | 64.3 | 63.2
  Week 12 [N=381,387] | 69.0 | 69.5
  Final visit [N=404,413] | 67.3 | 68.5
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.20, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.90 to 1.67]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.57, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.65 to 1.26]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.92, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.69 to 1.39]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.90, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.73 to 1.42]

17. Secondary Outcome: Change From Baseline to Week 4 in Mobility Scores as Assessed by the European Quality of Life 5-Dimensions (EQ-5D-5L) Questionnaire
Description: The European Quality of Life 5-Dimensions Questionnaire (EQ-5D-5L) is a standardized nondisease specific (i.e., generic) instrument for use as a measure of health outcome. It has 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each dimension has 5 response levels (e.g., no problems with performing activity, slight problems, moderate problems, severe problems, unable to perform [extreme problems]).
Time Frame: Baseline and Week 4
Population: FAS population who have non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 905 | 896
participants
  No problems -> No problems | 447 | 443
  No problems -> Slight problems | 45 | 43
  No problems -> Moderate problems | 23 | 19
  No problems -> Severe problems | 2 | 6
  No problems -> Extreme problems | 0 | 1
  No problems -> no data | 4 | 3
  Slight problems -> no problems | 66 | 80
  Slight problems -> slight problems | 47 | 47
  Slight problems -> moderate problems | 24 | 11
  Slight problems -> severe problems | 6 | 3
  Slight problems -> extreme problems | 0 | 1
  Slight problems -> no data | 1 | 1
  Moderate problems -> no problems | 39 | 51
  Moderate problems -> slight problems | 39 | 45
  Moderate problems -> moderate problems | 50 | 46
  Moderate problems -> severe problems | 7 | 6
  Moderate problems -> extreme problems | 1 | 0
  Moderate problems -> no data | 0 | 1
  Severe problems -> no problems | 20 | 16
  Severe problems -> slight problems | 24 | 34
  Severe problems -> moderate problems | 45 | 29
  Severe problems -> severe problems | 16 | 12
  Severe problems -> extreme problems | 1 | 0
  Severe problems -> no data | 0 | 2
  Extreme problems -> no problems | 2 | 1
  Extreme problems -> slight problems | 1 | 1
  Extreme problems -> moderate problems | 0 | 0
  Extreme problems -> severe problems | 0 | 0
  Extreme problems -> extreme problems | 0 | 1
  Extreme problems -> no data | 0 | 0
  No data -> no problems | 1 | 1
  No data -> slight problems | 1 | 1
  No data -> moderate problems | 1 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 8 | 7

18. Secondary Outcome: Change From Baseline to Week 4 in Self-care Scores as Assessed by the EQ-5D-5L Questionnaire
Description: The EQ-5D-5L is a standardized nondisease specific (i.e., generic) instrument for use as a measure of health outcome. It has 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each dimension has 5 response levels (e.g., no problems with performing activity, slight problems, moderate problems, severe problems, unable to perform [extreme problems]).
Time Frame: Baseline and Week 4
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 905 | 896
participants
  No problems -> No problems | 693 | 703
  No problems -> slight problems | 26 | 23
  No problems -> moderate problems | 12 | 4
  No problems -> severe problems | 0 | 0
  No problems -> extreme problems | 0 | 1
  No problems -> no data | 5 | 5
  Slight problems -> No problems | 37 | 41
  Slight problems -> slight problems | 28 | 16
  Slight problems -> moderate problems | 8 | 5
  Slight problems -> severe problems | 1 | 2
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 0 | 0
  Moderate problems -> no problems | 24 | 17
  Moderate problems -> slight problems | 18 | 28
  Moderate problems -> moderate problems | 17 | 15
  Moderate problems -> severe problems | 1 | 0
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 0 | 0
  Severe problems -> no problems | 9 | 15
  Severe problems -> slight problems | 13 | 15
  Severe problems -> moderate problems | 7 | 6
  Severe problems -> severe problems | 4 | 0
  Severe problems -> extreme problems | 0 | 1
  Severe problems -> no data | 0 | 1
  Extreme problems -> no problems | 4 | 1
  Extreme problems -> slight problems | 1 | 1
  Extreme problems -> moderate problems | 1 | 0
  Extreme problems -> severe problems | 0 | 2
  Extreme problems -> extreme problems | 1 | 0
  Extreme problems -> no data | 0 | 1
  No data -> no problems | 1 | 2
  No data -> slight problems | 1 | 0
  No data -> moderate problems | 1 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 8 | 7

19. Secondary Outcome: Change From Baseline to Week 4 in Usual Activities Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 4
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 905 | 896
participants
  No problems -> no problems | 421 | 422
  No problems -> slight problems | 61 | 63
  No problems -> moderate problems | 20 | 10
  No problems -> severe problems | 4 | 3
  No problems -> extreme problems | 1 | 0
  No problems -> no data | 4 | 4
  Slight problems -> no problems | 102 | 101
  Slight problems -> slight problems | 49 | 58
  Slight problems -> moderate problems | 14 | 16
  Slight problems -> severe problems | 2 | 1
  Slight problems -> extreme problems | 1 | 1
  Slight problems -> no data | 1 | 0
  Moderate problems -> no problems | 47 | 34
  Moderate problems -> slight problems | 59 | 59
  Moderate problems -> moderate problems | 45 | 39
  Moderate problems -> severe problems | 9 | 7
  Moderate problems -> extreme problems | 1 | 0
  Moderate problems -> no data | 0 | 0
  Severe problems -> no problems | 17 | 28
  Severe problems -> slight problems | 21 | 19
  Severe problems -> moderate problems | 11 | 13
  Severe problems -> severe problems | 7 | 7
  Severe problems -> extreme problems | 1 | 1
  Severe problems -> no data | 0 | 3
  Extreme problems -> no problems | 0 | 4
  Extreme problems -> slight problems | 3 | 5
  Extreme problems -> moderate problems | 5 | 3
  Extreme problems -> severe problems | 3 | 1
  Extreme problems -> extreme problems | 1 | 1
  Extreme problems -> no data | 0 | 0
  No data -> no problems | 0 | 2
  No data -> slight problems | 2 | 0
  No data -> moderate problems | 1 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 8 | 7

20. Secondary Outcome: Change From Baseline to Week 4 in Pain/Discomfort Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 4
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 905 | 896
participants
  No problems -> no problems | 299 | 285
  No problems -> slight problems | 57 | 67
  No problems -> moderate problems | 11 | 17
  No problems -> severe problems | 1 | 5
  No problems -> extreme problems | 1 | 0
  No problems -> no data | 2 | 4
  Slight problems -> no problems | 101 | 97
  Slight problems -> slight problems | 116 | 109
  Slight problems -> moderate problems | 32 | 25
  Slight problems -> severe problems | 2 | 4
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 1 | 0
  Moderate problems -> no problems | 51 | 44
  Moderate problems -> slight problems | 60 | 86
  Moderate problems -> moderate problems | 66 | 65
  Moderate problems -> severe problems | 10 | 12
  Moderate problems -> extrme problems | 1 | 1
  Moderate problems -> no data | 2 | 1
  Severe problems -> no problems | 21 | 19
  Severe problems -> slight problems | 22 | 25
  Severe problems -> moderate problems | 19 | 17
  Severe problems -> severe problems | 20 | 6
  Severe problems -> extreme problems | 6 | 0
  Severe problems -> no data | 0 | 1
  Extreme problems -> no problems | 1 | 1
  Extreme problems -> slight problems | 2 | 6
  Extreme problems -> moderate problems | 3 | 3
  Extreme problems -> severe problems | 1 | 2
  Extreme problems -> extreme problems | 2 | 0
  Extreme problems -> no data | 0 | 1
  No data -> no problems | 1 | 1
  No data -> slight problems | 0 | 1
  No data -> moderate problems | 2 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 8 | 7

21. Secondary Outcome: Change From Baseline to Week 4 in Anxiety/Depression Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 4
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 905 | 896
participants
  No problems -> no problems | 328 | 339
  No problems -> slight problems | 59 | 65
  No problems -> moderate problems | 11 | 11
  No problems -> severe problems | 2 | 2
  No problems -> extreme problems | 0 | 2
  No problems -> no data | 4 | 2
  Slight problems -> no problems | 98 | 102
  Slight problems -> slight problems | 122 | 94
  Slight problems -> moderate problems | 29 | 25
  Slight problems -> severe problems | 5 | 3
  Slight problems -> extreme problems | 1 | 0
  Slight problems -> no data | 0 | 0
  Moderate problems -> no problems | 25 | 33
  Moderate problems -> slight problems | 64 | 65
  Moderate problems -> moderate problems | 37 | 40
  Moderate problems -> severe problems | 12 | 10
  Moderate problems -> extreme problems | 3 | 1
  Moderate problems -> no data | 0 | 2
  Severe problems -> no problems | 12 | 17
  Severe problems -> slight problems | 32 | 29
  Severe problems -> moderate problems | 26 | 19
  Severe problems -> severe problems | 12 | 9
  Severe problems -> extreme problems | 2 | 0
  Severe problems -> no data | 1 | 3
  Extreme problems -> no problems | 7 | 12
  Extreme problems -> slight problems | 8 | 4
  Extreme problems -> moderate problems | 3 | 5
  Extreme problems -> severe problems | 4 | 4
  Extreme problems -> extreme problems | 3 | 5
  Extreme problems -> no data | 0 | 0
  No data -> no problems | 1 | 1
  No data -> slight problems | 2 | 1
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 8 | 7

22. Secondary Outcome: Change From Baseline to Week 8 in Mobility Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 8
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 882 | 875
participants
  No problems -> no problems | 445 | 446
  No problems -> slight problems | 38 | 31
  No problems -> moderate problems | 20 | 23
  No problems -> severe problems | 3 | 3
  No problems -> extreme problems | 1 | 1
  No problems -> no data | 14 | 11
  Slight problems -> no problems | 70 | 78
  Slight problems -> slight problems | 46 | 44
  Slight problems -> moderate problems | 19 | 12
  Slight problems -> severe problems | 3 | 3
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 6 | 6
  Moderate problems -> no problems | 51 | 47
  Moderate problems -> slight problems | 41 | 52
  Moderate problems -> modrate problems | 31 | 40
  Moderate problems -> severe problems | 8 | 6
  Moderate problems -> extreme problems | 1 | 0
  Moderate problems -> no data | 4 | 4
  Severe problems -> no problems | 30 | 22
  Severe problems -> slight problems | 30 | 41
  Severe problems -> moderate problems | 21 | 15
  Severe problems -> severe problems | 20 | 8
  Severe problems -> extreme problems | 1 | 0
  Severe problems -> no data | 4 | 7
  Extreme problems -> no problems | 1 | 0
  Extreme problems -> slight problems | 1 | 1
  Extreme problems -> moderate problems | 1 | 0
  Extreme problems -> severe problems | 0 | 1
  Extreme problems -> extreme problems | 0 | 1
  Extreme problems -> no data | 0 | 0
  No data -> no problems | 4 | 4
  No data -> slight problems | 3 | 1
  No data -> moderate problems | 1 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 3 | 4

23. Secondary Outcome: Change From Baseline to Week 8 in Self-care Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 8
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 882 | 875
participants
  No problems -> no problems | 672 | 673
  No problems -> slight problems | 35 | 38
  No problems -> moderate problems | 7 | 2
  No problems -> severe problems | 1 | 1
  No problems -> extreme problems | 1 | 1
  No problems -> no data | 20 | 21
  Slight problems -> no problems | 42 | 33
  Slight problems -> slight problems | 19 | 20
  Slight problems -> moderate problems | 9 | 9
  Slight problems -> severe problems | 1 | 0
  Slight problems -> exteme problems | 0 | 0
  Slight problems -> no data | 3 | 2
  Moderate problems -> no problems | 34 | 34
  Moderate problems -> slight problems | 17 | 16
  Moderate problems -> moderate problems | 5 | 6
  Moderate problems -> severe problems | 2 | 2
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 2 | 2
  Severe problems -> no problems | 17 | 13
  Severe problems -> slight problems | 9 | 15
  Severe problems -> moderate problems | 4 | 8
  Severe problems -> severe problems | 2 | 0
  Severe problems -> extreme problems | 0 | 0
  Severe problems -> no data | 1 | 2
  Extreme problems -> no problems | 1 | 2
  Extreme problems -> slight problems | 4 | 2
  Extreme problems -> moderate problems | 0 | 0
  Extreme problems -> severe problems | 0 | 0
  Extreme problems -> extreme problems | 0 | 0
  Extreme problems -> no data | 2 | 1
  No data -> no problems | 6 | 5
  No data -> slight problems | 2 | 0
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 3 | 4

24. Secondary Outcome: Change From Baseline to Week 8 in Usual Activities Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 8
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 882 | 875
participants
  No problems -> no problems | 430 | 426
  No problems -> slight problems | 48 | 49
  No problems -> moderate problems | 15 | 11
  No problems -> severe problems | 2 | 3
  No problems -> extreme problems | 0 | 0
  No problems -> no data | 16 | 13
  Slight problems -> no problems | 101 | 109
  Slight problems -> slight problems | 45 | 50
  Slight problems -> moderate problems | 16 | 12
  Slight problems -> severe problems | 3 | 2
  Slight problems -> extreme problems | 1 | 0
  Slight problems -> no data | 3 | 4
  Moderate problems -> no problems | 61 | 53
  Moderate problems -> slight problems | 57 | 53
  Moderate problems -> moderate problems | 26 | 20
  Moderate problems -> severe problems | 10 | 6
  Moderate problems -> extreme problems | 1 | 1
  Moderate problems -> no data | 6 | 6
  Severe problems -> no problems | 13 | 16
  Severe problems -> slight problems | 23 | 32
  Severe problems -> moderate problems | 12 | 15
  Severe problems -> severe problems | 7 | 3
  Severe problems -> extreme problems | 0 | 0
  Severe problems -> no data | 2 | 5
  Extreme problems -> no problems | 5 | 4
  Extreme problems -> slight problems | 2 | 5
  Extreme problems -> moderate problems | 2 | 3
  Extreme problems -> severe problems | 2 | 0
  Extreme problems -> extreme problems | 0 | 2
  Extreme problems -> no data | 1 | 0
  No data -> no problems | 3 | 4
  No data -> slight problems | 5 | 1
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 3 | 4

25. Secondary Outcome: Change From Baseline to Week 8 in Pain/Discomfort Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 8
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 882 | 875
participants
  No problems -> no problems | 291 | 286
  No problems -> slight problems | 52 | 66
  No problems -> moderate problems | 13 | 16
  No problems -> severe problems | 4 | 0
  No problems -> extreme problems | 1 | 0
  No problems -> no data | 10 | 10
  Slight problems -> no problems | 103 | 96
  Slight problems -> slight problems | 111 | 103
  Slight problems -> moderate problems | 25 | 30
  Slight problems -> severe problems | 6 | 1
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 7 | 5
  Moderate problems -> no problems | 59 | 61
  Moderate problems -> slight problems | 66 | 78
  Moderate problems -> moderate problems | 46 | 57
  Moderate problems -> severe problems | 10 | 4
  Moderate problems -> extreme problems | 1 | 1
  Moderate problems -> no data | 8 | 8
  Severe problems -> no problems | 17 | 16
  Severe problems -> slight problems | 37 | 25
  Severe problems -> moderate problems | 12 | 15
  Severe problems -> severe problems | 18 | 7
  Severe problems -> extreme problems | 2 | 1
  Severe problems -> no data | 2 | 4
  Extreme problems -> no problems | 1 | 3
  Extreme problems -> slight problems | 4 | 4
  Extreme problems -> moderate problems | 2 | 4
  Extreme problems -> severe problems | 0 | 1
  Extreme problems -> extreme problems | 1 | 0
  Extreme problems -> no data | 1 | 1
  No data -> no problems | 4 | 2
  No data -> slight problems | 4 | 3
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 3 | 4

26. Secondary Outcome: Change From Baseline to Week 8 in Anxiety/Depression Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 8
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 882 | 875
participants
  No problems -> no problems | 325 | 334
  No problems -> slight problems | 52 | 65
  No problems -> moderate problems | 15 | 8
  No problems -> severe problems | 2 | 1
  No problems -> extreme problems | 0 | 0
  No problems -> no data | 10 | 13
  Slight problems -> no problems | 122 | 116
  Slight problems -> slight problems | 94 | 79
  Slight problems -> moderate problems | 26 | 20
  Slight problems -> severe problems | 4 | 3
  Slight problems -> extreme problems | 3 | 2
  Slight problems -> no data | 6 | 4
  Moderate problems -> no problems | 42 | 49
  Moderate problems -> slight problems | 50 | 59
  Moderate problems -> moderate problems | 31 | 34
  Moderate problems -> severe problems | 11 | 4
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 7 | 5
  Severe problems -> no problems | 23 | 13
  Severe problems -> slight problems | 39 | 37
  Severe problems -> moderate problems | 11 | 12
  Severe problems -> severe problems | 7 | 6
  Severe problems -> extreme problems | 1 | 3
  Severe problems -> no data | 4 | 6
  Extreme problems -> no problems | 9 | 11
  Extreme problems -> slight problems | 7 | 10
  Extreme problems -> moderate problems | 2 | 4
  Extreme problems -> severe problems | 3 | 1
  Extreme problems -> extreme problems | 3 | 4
  Extreme problems -> no data | 1 | 0
  No data -> no problems | 5 | 2
  No data -> slight problems | 3 | 2
  No data -> moderate problems | 0 | 1
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 3 | 4

27. Secondary Outcome: Change From Baseline to Week 12 in Mobility Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 12
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 865 | 857
participants
  No problems -> no problems | 442 | 459
  No problems -> slight problems | 36 | 25
  No problems -> moderate problems | 10 | 10
  No problems -> severe problems | 6 | 5
  No problems -> extreme problems | 1 | 0
  No problems -> no data | 26 | 16
  Slight problems -> no problems | 77 | 82
  Slight problems -> slight problems | 43 | 32
  Slight problems -> moderate problems | 15 | 16
  Slight problems -> severe problems | 2 | 2
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 7 | 11
  Moderate problems -> no problems | 57 | 63
  Moderate problems -> slight problems | 31 | 43
  Moderate problems -> moderate problems | 35 | 30
  Moderate problems -> severe problems | 7 | 4
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 6 | 9
  Severe problems -> no problems | 53 | 51
  Severe problems -> slight problems | 15 | 17
  Severe problems -> moderate problems | 15 | 7
  Severe problems -> severe problems | 18 | 8
  Severe problems -> extreme problems | 0 | 0
  Severe problems -> no data | 5 | 10
  Extreme problems -> no problems | 2 | 1
  Extreme problems -> slight problems | 0 | 1
  Extreme problems -> moderate problems | 0 | 0
  Extreme problems -> severe problems | 0 | 0
  Extreme problems -> extreme problems | 0 | 1
  Extreme problems -> no data | 1 | 0
  No data -> no problems | 2 | 9
  No data -> slight problems | 5 | 0
  No data -> moderate problems | 3 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

28. Secondary Outcome: Change From Baseline to Week 12 in Self-care Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 12
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 865 | 857
participants
  No problems -> no problems | 667 | 670
  No problems -> slight problems | 26 | 23
  No problems -> moderate problems | 5 | 6
  No problems -> severe problems | 1 | 1
  No problems -> extreme problems | 1 | 0
  No problems -> no data | 36 | 36
  Slight problems -> no problems | 43 | 42
  Slight problems -> slight problems | 13 | 12
  Slight problems -> moderate problems | 14 | 5
  Slight problems -> severe problems | 1 | 1
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 3 | 4
  Moderate problems -> no problems | 44 | 46
  Moderate problems -> slight problems | 8 | 6
  Moderate problems -> moderate problems | 5 | 6
  Moderate problems -> severe problems | 1 | 0
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 2 | 2
  Severe problems -> no problems | 25 | 25
  Severe problems -> slight problems | 4 | 7
  Severe problems -> moderate problems | 0 | 2
  Severe problems -> severe problems | 3 | 1
  Severe problems -> extreme problems | 0 | 0
  Severe problems -> no data | 1 | 3
  Extreme problems -> no problems | 4 | 4
  Extreme problems -> slight problems | 0 | 0
  Extreme problems -> moderate problems | 0 | 0
  Extreme problems -> severe problems | 0 | 0
  Extreme problems -> extreme problems | 0 | 0
  Extreme problems -> no data | 3 | 1
  No data -> no problems | 8 | 9
  No data -> slight problems | 2 | 0
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

29. Secondary Outcome: Change From Baseline to Week 12 in Usual Activities Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 12
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 865 | 857
participants
  No problems -> no problems | 425 | 426
  No problems -> slight problems | 43 | 45
  No problems -> moderate problems | 14 | 7
  No problems -> severe problems | 2 | 2
  No problems -> extreme problems | 0 | 0
  No problems -> no data | 27 | 22
  Slight problems -> no problems | 103 | 107
  Slight problems -> slight problems | 45 | 53
  Slight problems -> moderate problems | 12 | 9
  Slight problems -> severe problems | 3 | 1
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 6 | 7
  Moderate problems -> no problems | 81 | 79
  Moderate problems -> slight problems | 41 | 31
  Moderate problems -> moderate problems | 25 | 15
  Moderate problems -> severe problems | 6 | 5
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 8 | 9
  Severe problems -> no problems | 31 | 40
  Severe problems -> slight problems | 7 | 13
  Severe problems -> moderate problems | 6 | 6
  Severe problems -> severe problems | 9 | 5
  Severe problems -> extreme problems | 1 | 0
  Severe problems -> no data | 3 | 7
  Extreme problems -> no problems | 7 | 7
  Extreme problems -> slight problems | 1 | 2
  Extreme problems -> moderate problems | 2 | 3
  Extreme problems -> severe problems | 1 | 1
  Extreme problems -> extreme problems | 0 | 0
  Extreme problems -> no data | 1 | 1
  No data -> no problems | 7 | 8
  No data -> slight problems | 3 | 1
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

30. Secondary Outcome: Change From Baseline to Week 12 in Pain/Discomfort Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 12
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 865 | 857
participants
  No problems -> no problems | 287 | 299
  No problems -> slight problems | 50 | 49
  No problems -> moderate problems | 15 | 11
  No problems -> severe problems | 2 | 4
  No problems -> extreme problems | 0 | 0
  No problems -> no data | 17 | 15
  Slight problems -> no problems | 112 | 116
  Slight problems -> slight problems | 97 | 87
  Slight problems -> moderate problems | 29 | 18
  Slight problems -> severe problems | 2 | 4
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 12 | 10
  Moderate problems -> no problems | 79 | 80
  Moderate problems -> slight problems | 49 | 71
  Moderate problems -> moderate problems | 42 | 38
  Moderate problems -> severe problems | 10 | 6
  Moderate problems -> extreme problems | 0 | 1
  Moderate problems -> no data | 10 | 13
  Severe problems -> no problems | 39 | 34
  Severe problems -> slight problems | 14 | 13
  Severe problems -> moderate problems | 16 | 12
  Severe problems -> severe problems | 12 | 1
  Severe problems -> extreme problems | 2 | 1
  Severe problems -> no data | 5 | 7
  Extreme problems -> no problems | 4 | 5
  Extreme problems -> slight problems | 2 | 2
  Extreme problems -> moderate problems | 1 | 3
  Extreme problems -> severe problems | 1 | 1
  Extreme problems -> extreme problems | 0 | 1
  Extreme problems -> no data | 1 | 1
  No data -> no problems | 7 | 5
  No data -> slight problems | 2 | 4
  No data -> moderate problems | 1 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

31. Secondary Outcome: Change From Baseline to Week 12 in Anxiety/Depression Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and Week 12
Population: FAS population who has non-missing values at both Baseline and specified visit.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 865 | 857
participants
  No problems -> no problems | 323 | 341
  No problems -> slight problems | 53 | 48
  No problems -> moderate problems | 10 | 10
  No problems -> severe problems | 1 | 2
  No problems -> extreme problems | 1 | 0
  No problems -> no data | 16 | 20
  Slight problems -> no problems | 132 | 118
  Slight problems -> slight problems | 84 | 80
  Slight problems -> moderate problems | 26 | 15
  Slight problems -> severe problems | 3 | 2
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 10 | 9
  Moderate problems -> no problems | 52 | 67
  Moderate problems -> slight problems | 51 | 44
  Moderate problems -> moderate problems | 18 | 28
  Moderate problems -> severe problems | 8 | 5
  Moderate problems -> extreme problems | 2 | 1
  Moderate problems -> no data | 10 | 6
  Severe problems -> no problems | 38 | 35
  Severe problems -> slight problems | 25 | 17
  Severe problems -> moderate problems | 7 | 14
  Severe problems -> severe problems | 9 | 2
  Severe problems -> extreme problems | 1 | 0
  Severe problems -> no data | 5 | 9
  Extreme problems -> no problems | 10 | 15
  Extreme problems -> slight problems | 5 | 2
  Extreme problems -> moderate problems | 3 | 7
  Extreme problems -> severe problems | 2 | 2
  Extreme problems -> extreme problems | 1 | 2
  Extreme problems -> no data | 4 | 2
  No data -> no problems | 9 | 7
  No data -> slight problems | 1 | 2
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

32. Secondary Outcome: Change From Baseline to Final Visit in Mobility Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and final visit (up to Week 12)
Population: FAS population who has non-missing values at both Baseline and specified visit. LOCF was used.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 906 | 897
participants
  No problems -> no problems | 460 | 471
  No problems -> slight problems | 37 | 25
  No problems -> moderate problems | 14 | 12
  No problems -> severe problems | 6 | 5
  No problems -> extreme problems | 1 | 0
  No problems -> no data | 3 | 2
  Slight problems -> no problems | 80 | 88
  Slight problems -> slight problems | 45 | 34
  Slight problems -> moderate problems | 16 | 18
  Slight problems -> severe problems | 2 | 2
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 1 | 1
  Moderate problems -> no problems | 60 | 67
  Moderate problems -> slight problems | 33 | 46
  Moderate problems -> moderate problems | 36 | 31
  Moderate problems -> severe problems | 7 | 4
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 0 | 1
  Severe problems -> no problems | 53 | 52
  Severe problems -> slight problems | 15 | 17
  Severe problems -> moderate problems | 17 | 11
  Severe problems -> severe problems | 20 | 11
  Severe problems -> extreme problems | 1 | 0
  Severe problems -> no data | 0 | 2
  Extreme problems -> no problems | 2 | 1
  Extreme problems -> slight problems | 1 | 1
  Extreme problems -> moderate problems | 0 | 0
  Extreme problems -> severe problems | 0 | 0
  Extreme problems -> extreme problems | 0 | 1
  Extreme problems -> no data | 0 | 0
  No data -> no problems | 2 | 9
  No data -> slight problems | 5 | 0
  No data -> moderate problems | 3 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

33. Secondary Outcome: Change From Baseline to Final Visit in Self-care Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and final visit (up to Week 12)
Population: FAS population who has non-missing values at both Baseline and specified visit. LOCF was used.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 906 | 897
participants
  No problems -> no problems | 697 | 699
  No problems -> slight problems | 27 | 26
  No problems -> moderate problems | 5 | 6
  No problems -> severe problems | 1 | 1
  No problems -> extreme problems | 2 | 0
  No problems -> no data | 4 | 4
  Slight problems -> no problems | 43 | 43
  Slight problems -> slight problems | 15 | 14
  Slight problems -> moderate problems | 15 | 6
  Slight problems -> severe problems | 1 | 1
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 0 | 0
  Moderate problems -> no problems | 45 | 46
  Moderate problems -> slight problems | 8 | 6
  Moderate problems -> moderate problems | 6 | 8
  Moderate problems -> severe problems | 1 | 0
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 0 | 0
  Severe problems -> no problems | 25 | 25
  Severe problems -> slight problems | 4 | 7
  Severe problems -> moderate problems | 0 | 4
  Severe problems -> severe problems | 4 | 1
  Severe problems -> extreme problems | 0 | 0
  Severe problems -> no data | 0 | 1
  Extreme problems -> no problems | 5 | 4
  Extreme problems -> slight problems | 1 | 0
  Extreme problems -> moderate problems | 0 | 0
  Extreme problems -> severe problems | 0 | 0
  Extreme problems -> extreme problems | 1 | 0
  Extreme problems -> no data | 0 | 1
  No data -> no problems | 8 | 9
  No data -> slight problems | 2 | 0
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme data | 0 | 0
  No data -> no data | 1 | 0

34. Secondary Outcome: Change From Baseline to Final Visit in Usual Activities Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and final visit (up to Week 12)
Population: FAS population who has non-missing values at both Baseline and specified visit. LOCF was used.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 906 | 897
participants
  No problems -> no problems | 444 | 440
  No problems -> slight problems | 46 | 49
  No problems -> moderate problems | 15 | 8
  No problems -> severe problems | 2 | 2
  No problems -> extreme problems | 0 | 0
  No problems -> no data | 4 | 3
  Slight problems -> no problems | 106 | 113
  Slight problems -> slight problems | 45 | 54
  Slight problems -> moderate problems | 15 | 9
  Slight problems -> severe problems | 3 | 1
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 0 | 0
  Moderate problems -> no problems | 83 | 79
  Moderate problems -> slight problems | 42 | 34
  Moderate problems -> moderate problems | 29 | 20
  Moderate problems -> severe problems | 7 | 6
  Moderate problems -> extreme problems | 0 | 0
  Moderate problems -> no data | 0 | 0
  Severe problems -> no problems | 31 | 41
  Severe problems -> slight problems | 9 | 14
  Severe problems -> moderate problems | 6 | 8
  Severe problems -> severe problems | 10 | 5
  Severe problems -> extreme problems | 1 | 0
  Severe problems -> no data | 0 | 3
  Extreme problems -> no problems | 7 | 7
  Extreme problems -> slight problem | 1 | 2
  Extreme problems -> moderate problem | 2 | 3
  Extreme problems -> severe problem | 1 | 1
  Extreme problems -> extreme problem | 1 | 1
  Extreme problems -> no data | 0 | 0
  No data -> no problems | 7 | 8
  No data -> slight problems | 3 | 1
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

35. Secondary Outcome: Change From Baseline to Final Visit in Pain/Discomfort Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and final visit (up to Week 12)
Population: FAS population who has non-missing values at both Baseline and specified visit. LOCF was used.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 906 | 897
participants
  No problems -> no problems | 297 | 306
  No problems -> slight problems | 55 | 52
  No problems -> moderate problems | 15 | 13
  No problems -> severe problems | 2 | 4
  No problems -> extreme problems | 0 | 0
  No problems -> no data | 2 | 3
  Slight problems -> no problems | 116 | 118
  Slight problems -> slight problems | 103 | 93
  Slight problems -> moderate problems | 30 | 20
  Slight problems -> severe problems | 2 | 4
  Slight problems -> extreme problems | 0 | 0
  Slight problems -> no data | 1 | 0
  Moderate problems -> no problems | 80 | 83
  Moderate problems -> slight problems | 51 | 72
  Moderate problems -> moderate problems | 48 | 44
  Moderate problems -> severe problems | 10 | 7
  Moderate problems -> extreme problems | 0 | 2
  Moderate problems -> no data | 1 | 1
  Severe problems -> no problems | 39 | 34
  Severe problems -> slight problems | 16 | 14
  Severe problems -> moderate problems | 16 | 15
  Severe problems -> severe problems | 15 | 3
  Severe problems -> extreme problems | 2 | 1
  Severe problems -> no data | 0 | 1
  Extreme problems -> no problems | 4 | 5
  Extreme problems -> slight problems | 2 | 2
  Extreme problems -> moderate problems | 1 | 3
  Extreme problems -> severe problems | 1 | 1
  Extreme problems -> extreme problems | 1 | 1
  Extreme problems -> no data | 0 | 1
  No data -> no problems | 7 | 5
  No data -> slight problems | 2 | 4
  No data -> moderate problems | 1 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

36. Secondary Outcome: Change From Baseline to Final Visit in Anxiety/Depression Scores as Assessed by the EQ-5D-5L Questionnaire
Description: as for outcome 18
Time Frame: Baseline and final visit (up to Week 12)
Population: FAS population who has non-missing values at both Baseline and specified visit. LOCF was used.
Measure: Number; unit: participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 906 | 897
participants
  No problems -> no problems | 332 | 356
  No problems -> slight problems | 55 | 52
  No problems -> moderate problems | 11 | 10
  No problems -> severe problems | 2 | 2
  No problems -> extreme problems | 1 | 0
  No problems -> no data | 3 | 1
  Slight problems -> no problems | 133 | 121
  Slight problems -> slight problems | 92 | 83
  Slight problems -> moderate problems | 26 | 17
  Slight problems -> severe problems | 4 | 2
  Slight problems -> extreme problems | 0 | 1
  Slight problems -> no data | 0 | 0
  Moderate problems -> no problems | 55 | 68
  Moderate problems -> slight problems | 52 | 45
  Moderate problems -> moderate problems | 22 | 29
  Moderate problems -> severe problems | 10 | 6
  Moderate problems -> extreme problems | 2 | 1
  Moderate problems -> no data | 0 | 2
  Severe problems -> no problems | 38 | 35
  Severe problems -> slight problems | 25 | 18
  Severe problems -> moderate problems | 8 | 15
  Severe problems -> severe problems | 12 | 6
  Severe problems -> extreme problems | 1 | 0
  Severe problems -> no data | 1 | 3
  Extreme problems -> no problems | 10 | 15
  Extreme problems -> slight problems | 6 | 2
  Extreme problems -> moderate problems | 3 | 7
  Extreme problems -> severe problems | 3 | 3
  Extreme problems -> extreme problems | 3 | 3
  Extreme problems -> no data | 0 | 0
  No data -> no problems | 9 | 7
  No data -> slight problems | 1 | 2
  No data -> moderate problems | 0 | 0
  No data -> severe problems | 0 | 0
  No data -> extreme problems | 0 | 0
  No data -> no data | 1 | 0

37. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12, and at the Final Visit in Symptom Bother Score as Assessed by the Overactive Bladder Questionnaire (OAB-q)
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to symptom bother and health-related quality of life (HRQoL). The symptom bother portion consists of 8 items, scored from 1 to 6. The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). A negative change from baseline indicates an improvement.
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: FAS population. LOCF was used for final visit only. N is the number of participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
units on a scale
  Week 4 [N=905,896] | -20.51 (0.576) | -22.20 (0.579)
  Week 8 [N=882,875] | -25.96 (0.599) | -27.76 (0.601)
  Week 12 [N=865,859] | -29.74 (0.647) | -31.84 (0.649)
  Final visit [N=906,897] | -28.89 (0.652) | -30.76 (0.655)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 4 Difference vs. Mirabegron. Difference of the adjusted mean is calculated by subtracting the adjusted mean of mirabegron from the adjusted mean of solifenacin; Test type: Superiority or Other; p = 0.039, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; Treatment group, gender, age group (<65, ≥65), number of prior antimuscarinics (1, ≥2), geographic region as fixed factors and baseline as covariate; Least squares mean difference = -1.69, 95% CI 2-sided [-3.29 to -0.08], Standard Error of Mean 0.817
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 8 Difference vs. Mirabegron. Difference of the adjusted mean is calculated by subtracting the adjusted mean of mirabegron from the adjusted mean of solifenacin; Test type: Superiority or Other; p = 0.034, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = -1.80, 95% CI 2-sided [-3.46 to -0.13], Standard Error of Mean 0.849
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.022, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = -2.10, 95% CI 2-sided [-3.90 to -0.30], Standard Error of Mean 0.917
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final Visit Difference vs. Mirabegron. Difference of the adjusted mean is calculated by subtracting the adjusted mean of mirabegron from the adjusted mean of solifenacin; Test type: Superiority or Other; p = 0.043, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = -1.87, 95% CI 2-sided [-3.68 to -0.06], Standard Error of Mean 0.924

38. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12, and at the Final Visit in Total Health-Related Quality of Life (HRQoL) Score as Assessed by the OAB-q
Description: The OAB-q is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: coping, concern, sleep, social interaction). The total score is calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: as for outcome 37
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
units on a scale
  Week 4 [N=905,896] | 17.09 (0.543) | 18.23 (0.546)
  Week 8 [N=882,875] | 21.66 (0.568) | 23.20 (0.570)
  Week 12 [N=865,859] | 25.31 (0.611) | 26.85 (0.613)
  Final visit [N=906,897] | 24.53 (0.616) | 25.94 (0.619)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 37, analysis 1]; Test type: Superiority or Other; p = 0.14, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = 1.14, 95% CI 2-sided [-0.37 to 2.65], Standard Error of Mean 0.770
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 37, analysis 2]; Test type: Superiority or Other; p = 0.055, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; Treatment group, gender, age group (<65, ≥65), number of prior antimuscarinics (1, ≥2), geographic region as fixed factors and baseline as covariates; Least squares mean difference = 1.55, 95% CI 2-sided [-0.03 to 3.13], Standard Error of Mean 0.805
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.074, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 38, analysis 2]; Least squares mean difference = 1.55, 95% CI 2-sided [-0.15 to 3.25], Standard Error of Mean 0.866
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 37, analysis 4]; Test type: Superiority or Other; p = 0.11, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 38, analysis 2]; Least squares mean difference = 1.41, 95% CI 2-sided [-0.30 to 3.12], Standard Error of Mean 0.873

39. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12, and at the Final Visit in Patient Perception of Bladder Condition (PPBC)
Description: The Patient Perception of Bladder Condition (PPBC) questionnaire is a single-item questionnare used to assess participants' perceptions and impressions of their bladder condition. Participants assessed their bladder condition using a 6-point categorical scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems.
Time Frame: Baseline and Week 4, Week 8, Week 12
Population: as for outcome 37
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
units on a scale
  Week 4 [N=905,896] | -0.91 (0.035) | -1.00 (0.035)
  Week 8 [N=882,875] | -1.30 (0.038) | -1.46 (0.038)
  Week 12 [N=865,858] | -1.58 (0.042) | -1.73 (0.042)
  Final visit [N=906,897] | -1.53 (0.042) | -1.67 (0.042)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 37, analysis 1]; Test type: Superiority or Other; p = 0.070, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = -0.09, 95% CI 2-sided [-0.19 to 0.01], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 37, analysis 2]; Test type: Superiority or Other; p = 0.003, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = -0.16, 95% CI 2-sided [-0.27 to -0.06], Standard Error of Mean 0.054
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Difference vs. Mirabegron.Difference of the adjusted mean is calculated by subtracting the adjusted mean of mirabegron from the adjusted mean of solifenacin; Test type: Superiority or Other; p = 0.015, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = -0.15, 95% CI 2-sided [-0.26 to -0.03], Standard Error of Mean 0.060
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 37, analysis 4]; Test type: Superiority or Other; p = 0.021, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = -0.14, 95% CI 2-sided [-0.25 to -0.02], Standard Error of Mean 0.059

40. Secondary Outcome: Change From Baseline to Week 12 and the Final Visit in the Patient's Assessment of Treatment Satisfaction (TS)-Visual Analog Scale (VAS)
Description: The Treatment Satisfaction (TS)-Visual Analogue Scale (VAS) was a self-rated scale with the participant answering the question "Are you satisfied with your treatment?" and placing a vertical mark on a line from 0 (No, not at all) to 10 (Yes, completely).
Time Frame: Baseline and Week 12
Population: as for outcome 37
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
units on a scale
  Week 12 [N=865,857] | 3.51 (0.099) | 3.93 (0.100)
  Final visit [N=891,876] | 3.44 (0.099) | 3.86 (0.100)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.002, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = 0.43, 95% CI 2-sided [0.15 to 0.70], Standard Error of Mean 0.141
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 37, analysis 4]; Test type: Superiority or Other; p = 0.003, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = 0.42, 95% CI 2-sided [0.14 to 0.70], Standard Error of Mean 0.141

41. Secondary Outcome: Change From Baseline to Week 12 and the Final Visit in the Patient's Assessment of Treatment Satisfaction Questionnaire-Likert Scale
Description: The Treatment Satisfaction (TS)-Likert Scale was a self-rated scale with the participant answering the question "How satisfied were you with your treatment?" with on a scale from 1 (extremely dissatisfied) to 7 (extremely satisfied).
Time Frame: Baseline and Week 12
Population: as for outcome 37
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
units on a scale
  Week 12 [N=876,871] | 2.92 (0.050) | 3.07 (0.050)
  Final visit [N=897,889] | 2.88 (0.050) | 3.03 (0.050)
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.027, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean diffrence = 0.16, 95% CI 2-sided [0.02 to 0.29], Standard Error of Mean 0.070
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; [analysis description as in outcome 37, analysis 4]; Test type: Superiority or Other; p = 0.034, ANCOVA — If p<0.05, this indicates superiority in favor of the treatment group with the largest improvement at specified visit; [statistical method as in outcome 37, analysis 1]; Least squares mean difference = 0.15, 95% CI 2-sided [0.01 to 0.29], Standard Error of Mean 0.071

42. Secondary Outcome: Percentage of Participants With Improvement in Symptom Bother Score as Assessed by the OAB-q: ≥ 10 Points Improvement in OAB-q at Week 12 and Final Visit
Description: A responder is defined as a participant with ≥10 points improvement in symptom bother from baseline.
Time Frame: Baseline to Week 12
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
percentage of participants
  Week 12 [N=865,859] | 77.5 | 82.4
  Final visit [N=906,897] | 76.2 | 81.2
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.010, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Treatment group, gender, age group (<65, ≥65), number of prior antimuscarinics (1, ≥2), geographic region and baseline value as factors; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.08 to 1.81]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.011, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.07 to 1.75]

43. Secondary Outcome: Percentage of Participants With Improvement in HRQoL Scales as Assessed by the OAB-q: ≥10 Points Improvement in OAB-q at Week 12 and Final Visit
Description: A responder is defined as a participant with >=10 points improvement in the total HRQL score from baseline.
Time Frame: Baseline to Week 12
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
percentage of participants
  Week 12 [N=865,859] | 69.2 | 72.6
  Final visit [N=906,897] | 67.5 | 71.0
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.037, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.28, 95% CI 2-sided [1.02 to 1.62]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.045, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.01 to 1.57]

44. Secondary Outcome: Percentage of Participants With Improvement of Treatment Satisfaction Questionnaire - Likert Scale: ≥1, ≥2, ≥3, ≥4, ≥5, and 6-point Improvement From Baseline to Week 12
Description: A responder is defined as a participant with ≥1, ≥2, ≥3, ≥4, ≥5 or 6-point improvement from baseline in TS-Likert scale.
Time Frame: Baseline to Week 12
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 876 | 871
percentage of participants
  ≥1 point improvement | 86.4 | 90.4
  ≥2 point improvement | 80.3 | 83.6
  ≥3 point improvement | 67.7 | 71.9
  ≥4 point improvement | 44.4 | 47.5
  ≥5 point improvement | 15.6 | 15.4
  6 point improvement | 2.5 | 2.9
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 (≥1 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.009, Regression, Logistic — Iif p<0.05, this indicates superiority in favor of the treatment group with the largest percentage of responders at specified visit; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.11 to 2.06]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 (≥2 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.065, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.99 to 1.65]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 (≥3 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.051, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.00 to 1.55]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 (≥4 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.14, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.95 to 1.47]
Statistical Analysis 5: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 (≥5 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.89, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.75 to 1.40]
Statistical Analysis 6: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 (6 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.66, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.64 to 2.04] — Participants from Canada were therefore excluded from this analysis due to low participant numbers

45. Secondary Outcome: Percentage of Participants With Improvement in Treatment Satisfaction Questionnaire - Likert Scale: ≥1, ≥2, ≥3, ≥4, ≥5, and 6-point Improvement From Baseline to Final Visit
Description: A responder is defined as a participant with >=1 or >=2 or >=3 or >=4 or >=5 or 6-point improvement from baseline in TS-Likert scale.
Time Frame: Baseline to final visit (up to Week 12)
Population: FAS population. LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 897 | 889
percentage of participants
  ≥1 point improvement | 85.6 | 89.4
  ≥2 point improvement | 79.0 | 82.6
  ≥3 point improvement | 66.7 | 70.8
  ≥4 point improvement | 43.8 | 46.6
  ≥5 point improvement | 15.4 | 15.1
  6 point improvement | 2.5 | 2.8
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit (≥1 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.016, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.07 to 1.93]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit (≥2 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.063, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.99 to 1.62]
Statistical Analysis 3: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit (≥3 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.054, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [1.00 to 1.53]
Statistical Analysis 4: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit (≥4 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.15, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.95 to 1.46]
Statistical Analysis 5: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit (≥5 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.75, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.77 to 1.44]
Statistical Analysis 6: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit (6 point improvement) Odds Rato vs. Mirabegron; Test type: Superiority or Other; p = 0.66, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.64 to 2.04] — Participants from Canada were therefore excluded from this analysis due to low participant numbers

46. Secondary Outcome: Percentage of Participants With Improvement in PPBC: ≥1 Point Improvement at Week 12 and Final Visit
Description: A responder is defined as a participant with ≥1 point improvement in PPBC from baseline.
Time Frame: Baseline to Week 12
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
percentage of participants
  Week 12 [N=865,858] | 73.1 | 76.7
  Final visit [N=906,897] | 71.9 | 74.9
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.082, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.97 to 1.57]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.15, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.94 to 1.49]

47. Secondary Outcome: Percentage of Participants With Major Improvement in PPBC: ≥2 Point Improvement at Week 12 and Final Visit
Description: A responder is defined as a participant with ≥2 point improvement in PPBC from baseline.
Time Frame: Baseline to Week 12
Population: as for outcome 37
Measure: Number; unit: percentage of participants
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Number analyzed (Participants) | 921 | 912
percentage of participants
  Week 12 [N=865,858] | 47.6 | 52.6
  Final visit [N=906,897] | 46.2 | 51.1
Statistical Analysis 1: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Week 12 Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.058, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.99 to 1.53]
Statistical Analysis 2: Comparison: Mirabegron 50 mg vs Solifenacin 5 mg; Final visit Odds Ratio vs. Mirabegron; Test type: Superiority or Other; p = 0.069, Regression, Logistic — If p<0.05, this indicates superiority in favor of the treatment group with the largest percentage of responders at specified visitI; [statistical method as in outcome 42, analysis 1]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.99 to 1.50]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 16 weeks)
Description: Safety Analysis Set population
Arm/Group | Mirabegron 50 mg | Solifenacin 5 mg
Serious Adverse Events (participants affected / at risk) | 14/936 | 13/934
Other Adverse Events (participants affected / at risk) | 29/936 | 54/934
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron 50 mg (N=936) | Solifenacin 5 mg (N=934)
Pneumonia (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Open angle glaucoma (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Dysplasia (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirabegron 50 mg (N=936) | Solifenacin 5 mg (N=934)
Dry mouth (Gastrointestinal disorders) | 29 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript 45 days prior to publication for review and comment.

Sponsor may delay the publication to seek patent protection.